CLINICAL TRIAL: NCT06701370
Title: The Effect of Task-oriented Training With Conventional Rehabilitation on Upper Extremity Motor Functions in Chronic Stroke Patients
Brief Title: The Effect of Task-oriented Training on Upper Extremity Motor Functions in Chronic Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biruni University (Other)
Responsible Party: Principal Investigator, Guzin Kaya Aytutuldu, Assist.Prof.Dr., Biruni University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BiruniUnive.
Record Dates: First submitted 2024-11-20; First posted 2024-11-22 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Stroke Patients; Chronic Stroke Patients
Keywords: task oriented training, stroke, exercise, upper extremity
MeSH Terms: conditions — Stroke; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Task oriented Training Group (Experimental): Conventional rehabilitation + Upper arm Ergometer
  + Task oriented Training
  Interventions: Other: Task Oriented Training; Other: Conventional Rehabilitation; Other: Upper arm ergometer
- Conventional Rehabilitation Group (Active Comparator): Conventional rehabilitation + Upper arm Ergometer
  Interventions: Other: Conventional Rehabilitation; Other: Upper arm ergometer

INTERVENTIONS:
Other: Task Oriented Training — Task oriented training consists of opening the bottlecap, stacking cubes on different sizes, buttoning,screwing, wearing a coat.
  Arms: Task oriented Training Group
Other: Conventional Rehabilitation — Bobath weightbearing and mobility exercises for upper extremity and 15 minutes Neuromuscular Electrical Stimulation.
Other: Upper arm ergometer — The patients will be rode 5 minutes forwardly and 5 minutes backwardly

SUMMARY:
The aim of our study was to investigate the effects of task-oriented training added to conventional rehabilitation on upper extremity muscle thickness and upper extremity motor functions.

DETAILED DESCRIPTION:
Stroke refers to a neurological disorder caused by cerebrovascular damage. It is defined as a sudden brain attack that causes partial or complete brain dysfunction due to blockage or rupture of blood vessels of the brain.The primary symptom of stroke is hemiparesis. In addition, stroke negatively affects senses, motor function, perception, cognition and language, depending on location, etiology and infarct volume. One study reported that %85 of stroke patients had hemiparesis and more than %69 had upper limp disfunction. In general, upper limb dysfunction not only causes problem in performing tasks that require fine motor skills (Daily tasks such as personal hygiene activities, eating and handwriting), but also makes ıt very difficult the perform tasks that require gross motor skills (such as balancing).(walking and self protection reflexes). Upper limb dysfunction reduces the quality of life (QoL) of patients with paralysis. It limits their ability to live independently in society as it impairs many of the basic IADLs (such as crawling, balancing, walking, writing, eating, washing and manipulating objects) necessary for individuals to live independently. Hands and arms are used in a wide range of tasks performed in the workplace and used to communicate.They also play an important role in various cognitive activities and motor functions. In stroke patients, the recovery of upper limb function, which is necessary to independently perform IADLs, can be considered as critical as the recovery of walking. The aim of therapeutic training in rehabilitation is to help patients try to use the affected side and voluntarily perform motor functions, and there are various physical intervention approaches.According to several recent studies conducted in stroke patients, among them, task-oriented training is reported to be effective in developing functional motor skills necessary to perform activities of daily living. Task-oriented training can help patients to increase their ability to perform IADLs. Training consists of a variety of functional activities that offer a more effective treatment approach. Task-oriented training is a therapeutic model based on the theory of motor control system, which regulates the movements of organisms by the nervous system, including reflexes. It uses a functional approach in the rehabilitation of neurological patients and teaches patients task-specific strategies to help them adapt to changing environments. The approach involves patients practicing a skill necessary to achieve the goal of a task to facilitate problem solving by improving their ability to adapt to various situations and developing an effective reward strategy. In addition, the approach for maximal learning involves motivating patients behaviorally using tasks related to their personal daily lives and emphasizes the interaction between patients and their environment. Task-focused training uses a patient-centered approach rather than a therapist-centered approach, and meaningful tasks are selected as a core component. The therapeutic goal of task-focused training is maximal recovery of motor function through proactive performance of activities using the upper limb on the affected side rather than the intact side . It was stated that repetitive and focused task-oriented training improves recovery of upper limb function and can improve motor order, dexterity and agility in the upper limb.

Lee also reported that task-oriented circuit training improved upper limb functions, performance in activities of daily living, and self-efficacy in expressing confidence.

The aim of our study was to investigate the effects of task-oriented training added to conventional rehabilitation on upper extremity muscle thickness and upper extremity motor functions.

ELIGIBILITY:
Inclusion Criteria:

* History of cerebrovascular accident at least 6 months ago;
* Score at least 20 points on the mini mental test;
* Not having pain with tension or severe weakness in the shoulder muscles;
* Active shoulder flexion movement of at least 30 degrees
* Having a stroke for the first time
* The level of motor function is Stage 3 or Stage 4 in Brunnstrom Staging according to the proximal function of the upper extremity
* Not receiving botulinum toxin treatment for the last 3 months

Exclusion Criteria:

* Presence of concomitant neurological, orthopedic, cardiovascular diseases and severe comorbidities
* Severe spasticity of the elbow flexors more than 2 on the Modified Ashworth Scale

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2024-10-30 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2025-03-30 (Actual)

PRIMARY OUTCOMES:
Fugl Meyer Upper extremity assessment | 5 minutes
  It is a disease-specific, objective motor impairment scale designed especially for the evaluation of recovery in hemiplegic patients after stroke. It includes subsections evaluating joint movements, coordination and reflex activities related to the shoulder, elbow, forearm, wrist and hand. The highest score that can be obtained from this assessment is 66. The assessment is applied to the affected upper extremities of individuals in the sitting position. The evaluated joint movements are scored as 0: no movement, 1: partial movement and 2: normal movement. Reflex activity is assessed using a reflex hammer and scored as 0: no reflex activity, 2: reflex activity can be elicited.
Wolf Motor Function Scale | 5 minutes
  It is an assessment method developed to evaluate motor skills and used in patients with moderate to severe upper extremity motor deficits. The original version was developed by Wolf et al. The modified version was used in our study and the validity and internal consistency of the WMFT have been proven. The test includes 17 activities. For 15 of the 17 activities, data are collected in two areas: "Functional Skill" and 'Performance Time". The other 2 activities evaluating muscle strength were not used in our study. The duration of the test is 30-45 minutes. Each activity was scored by the physiotherapist on a 0-5 point scale (0= Never used the affected hand during the activity, 5= Normal movement) using the "Functional skill scale". An average score should be calculated for the functional skills scale. Accordingly, the patient can score between 0-5 points in this evaluation and a high score indicates good functional skills. "Performance Time" is recorded in seconds. The
Examination of muscle thickness by ultrasound | 10 minutes
  Muscle thickness of the biceps, triceps and anterior deltoid muscles on the hemiplegic and intact side will be measured and recorded by ultrosound before and after treatment.

SECONDARY OUTCOMES:
Motor Activity Log-28 | 5 minutes
  MAG-28 is a structured assessment designed to examine how often and how well the person uses the affected arm outside the treatment session. The reason for choosing the 28-activity form of MAG, which can be found in many forms in the literature such as MAG-14 and MAG-30, in our study is that its validity and reliability have been proven. MAG-28 consists of two scales that question how often the patient uses the upper extremity of the affected side for each activity (Frequency of Use Scale) and how well the patient can perform the activity (Movement Quality Scale) during 28 daily activities (turning on a light switch, opening a door, etc.). The scales are printed on separate sheets of paper and remain in front of the patient being assessed throughout the administration of the test.
2 minutes walking test | 5 minutes
  The test protocol will follow the guidelines recommended by Pin (24). The 2-minute walk test is repeated 2 times with a 10-minute rest between each trial to minimize fatigue in individuals. Each individual sits in a chair for 10 minutes before the 2-minute walk test. Each individual is asked to walk at their own pace without running for 2 minutes on a quiet, 10 m long concrete walkway. The start and end points of the walkway are clearly marked with brightly colored marker tape. Individuals are allowed to rest or stop at any time during the 2 minutes if necessary.
Grip strength | 3 minutes
  Hand grip strength of the patients will be measured with Jamar Hand Dynamometer. The Jamar Hand Dynamometer has 5 different handles that can be adapted according to the patient's hand size . For the measurement, the patients are seated and the elbow is flexed ninety degrees, the forearm is in neutral position and the wrist is in extension between zero and thirty degrees. Measurements were taken for both sides and three measurements were taken at thirty-sixty second intervals and the average of the three measurements was recorded.
Functional Independence Measurements | 10 minutes
  Defined as a comprehensive scale, the FIM assesses the functions of the individual in two main areas evaluates:
  1. Physical/motor functions (13 items)
  2. Cognitive functions (5 items) The items are a seven-level scale assessing different activities such as self-care, sphincter control, transfer, locomotion, communication and social perception. Level 1: Complete Dependence, Level 7: Complete Independence. The FIM total score is obtained by summing the scores of the 18 items. The maximum score can be 126 and the minimum score can be 18. A high total score indicates that the individual's dependence in Activities of Daily Living (ADL) decreases . Functional Independence Scale is presented in Appendix-8. All items should be evaluated and not left blank. Items are evaluated by sticking to the activities defined. For example, when questioning sphincter control, going to the toilet or sitting on the toilet is not taken into consideration.

CONTACTS AND LOCATIONS:
Locations (1):
- Biruni University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
We share it in order to contribute to future studies.
Supporting Information: Study Protocol, SAP
Time Frame: september 30- march 30

REFERENCES:
- [Result] Chang JJ, Tung WL, Wu WL, Su FC. Effect of bilateral reaching on affected arm motor control in stroke--with and without loading on unaffected arm. Disabil Rehabil. 2006 Dec 30;28(24):1507-16. doi: 10.1080/09638280600646060. PMID 17178614
- [Result] Yoo DH, Kim SY. Effects of upper limb robot-assisted therapy in the rehabilitation of stroke patients. J Phys Ther Sci. 2015 Mar;27(3):677-9. doi: 10.1589/jpts.27.677. Epub 2015 Mar 31. PMID 25931706
- [Result] Michaelsen SM, Dannenbaum R, Levin MF. Task-specific training with trunk restraint on arm recovery in stroke: randomized control trial. Stroke. 2006 Jan;37(1):186-92. doi: 10.1161/01.STR.0000196940.20446.c9. Epub 2005 Dec 8. PMID 16339469